CLINICAL TRIAL: NCT02333006
Title: Anosognosia Evaluation After Cranocerebral Trauma Moderate to Severe
Acronym: ANOSOGNOSIA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Responsible Party: Principal Investigator, AZOUVI, MDPHD, Centre d'Investigation Clinique et Technologique 805
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2014-A00110-47
Record Dates: First submitted 2014-12-24; First posted 2015-01-07 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Traumatic Brain Injury
Keywords: Anosognosia
MeSH Terms: conditions — Brain Injuries, Traumatic; Agnosia | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Traumatic brain injury questionnaires (Other): Traumatic brain injury patients with anosognosia will answer to quetionnaires about Anosognosia compare to the answer of participant without neurological deficits
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Traumatic brain injury patients and participant without neurological deficits will answer to questionnaires about Anosognosia

SUMMARY:
This study is conducted over 18 months. The main objective of this study is to test and compare the relevance and reliability of different tools for measuring the anosognosia.

Secondary objectives are :

* identify the relevant test who are able to evaluate more specially the cognitive processes involved in anosognosia
* explore the links between the anosognosia manifestations and the psychological manifestations

DETAILED DESCRIPTION:
This experimental protocol is proposed to 40 patients who have a moderate or severe traumatic brain injury. All of this protocol is 2 hours, tasks are administered in the order named.

To measure anosognosia, this protocol is to administer 4 questionnaires used in clinical routine who have proposed to patients and their therapist and relative who know them well. The chosen measure is the difference between the results of the patient and that of the therapist or relative. Others evaluations are administrated to question the beliefs capacity during 2 certainty of judgment tasks replicated or adapted articles from the literature (tasks of guessing and task of judgments facts).

The patients are also evaluated through several executive tasks (who come from battery of tests called 'Groupe de Reflexion sur l'évaluation des fonctions exécutives') and global cognitive efficiency tasks from the Wechsler Adult Intelligence Scale (involving non-verbal reasoning, psychomotor speed and general knowledge). These different tests measure the capacity of inhibition, mental flexibility, planning and information generation.

At last, mood and coping strategy questionnaires are proposed to patients for complete this protocol.

This protocol are also administered to 40 volunteers who have not had traumatic brain injury to monitor standards in general population (because all these tasks are not systematically standardized).

ELIGIBILITY:
Inclusion Criteria:

* patients with a moderate or severe traumatic brain injury occurred at least 3 months ago (Glasgow ≤ 12 or duration of post-traumatic amnesia > 1 week)
* patients ≥ 18 years old and who have signed a letter of information

Exclusion Criteria :

* motor, sensitive and phasic disorders who are not allowing the test passation
* neurological or psychiatric antecedents
* patients who refused to participate in the study
* non affiliation to a social security scheme
* patients under guardianship or trusteeship

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-02; Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Anosognosia score | 1h30
  Questionaire about anosognosia

SECONDARY OUTCOMES:
Neuropsychological score | 1h
  Neuropsychological tests

CONTACTS AND LOCATIONS:
Overall Officials: EMILIE DROMER, Psychologue, Study Chair — Raymond Poincaré Hospital
Locations (1):
- Hopital Raymond Poincare, Garches, France